CLINICAL TRIAL: NCT05502029
Title: Translating Anesthetic Care Throughout: A Feasibility Randomized Trial
Brief Title: Translating Anesthesia Care Throughout
Acronym: TACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mount Zion Health Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22-36587
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Limited English Proficiency; Perioperative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Translator in preoperative area
  Interventions: Behavioral: Standard translation
- Intervention (Experimental): Translator in preoperative area, continued through transport to the operating room, and in the operating room until the patient is under general anesthesia
  Interventions: Behavioral: Extended translation

INTERVENTIONS:
Behavioral: Extended translation — Translation extended beyond the preoperative area
  Arms: Intervention
Behavioral: Standard translation — Translation in the preoperative area
  Arms: Control

SUMMARY:
Patients with limited English proficiency (LEP) are at significant risk of receiving care different from those who are English proficient. Through Translating Anesthetic Care Throughout (TACT), the investigators aim to reduce the disparities experienced by participants with LEP undergoing anesthesia by continuing language translation from the preoperative area into the operating room, where participants will be better able to understand what is happening in an otherwise foreign environment. At this time, some participants receive translation in the preoperative area using an interpreter. No further translation is provided beyond the preoperative area unless there is a provider with language concordance or interpretation skills within the perioperative team. The investigators plan to study how extended translation changes a participant's understanding of and feelings about the perioperative period. Supporting language translation for LEP participants from the preoperative area into their operating room (OR) experience will enable providers to better understand how to care for participants from different cultural and language backgrounds and will help us understand how to better serve our community at large. The investigators hypothesize that participants who receive continual translation will have improved informed consent, have improved trust of their anesthesia providers, and be more satisfied with patient care. In addition, they anticipate that the care team also will benefit by the enhanced communication with the participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants who identify another language other than English as their preferred language
* Participants with planned general anesthesia

Exclusion Criteria:

* Participants whose preferred language is documented as English
* Participants with planned sedation or monitored anesthesia care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Informed consent success as assessed by Likert scale | One week after general anesthesia
  The participant will be asked how well their anesthesia provider prepared them for their general anesthesia experience. A 5-point Likert scale response will be used for the assessment ranging from 1 (not at all) to 5 (extremely well).
Participant trust as assessed by survey | One week after general anesthesia
  Participants will be asked whether they trusted their provider(s) using a yes/no response.
Participant satisfaction as assessed by Likert scale | One week after general anesthesia
  Participants will be asked whether they were satisfied with their anesthesia experience using a yes/no response.

SECONDARY OUTCOMES:
Participant anxiety as assessed by the Amsterdam Preoperative Anxiety and Information Scale | The day before surgery
  The Amsterdam Preoperative Anxiety and Information Scale (APAIS) is a 6-question validated tool used to generate a score to assess a patient's level of preoperative anxiety. Questions 1, 2, 4, and 5 represent anxiety. Each of these questions is assessed with a Likert scale in which 1 rpresents agreement of not at all and 5 represents extremely. Scores from the four anxiety-representing questions are totaled with a possible range from 4 to 20 with a lower score indicating less anxiety and a higher score more anxiety. A score of greater than or equal to 11 signifies participant anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Odmara Barreto Chang, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center at Mount Zion, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study whose results are intended to inform the investigators of whether additional study is warranted.